CLINICAL TRIAL: NCT01950780
Title: An Open-Label Pilot Study to Evaluate the Efficacy of Ruxolitinib in Moderate to Severe Alopecia Areata
Brief Title: Pilot Study to Evaluate the Efficacy of Ruxolitinib in Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Locks of Love (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAL7102
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Ruxolitinib
MeSH Terms: conditions — Alopecia Areata | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib (Experimental): A fixed dose of ruxolitinib (20mg) will be self-administered orally twice daily for 12 to 24 weeks. Dosing may be decreased or held if needed due to adverse effects.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — A fixed dose of ruxolitinib (20mg) will be self-administered orally twice daily for 12 to 24 weeks. Dosing may be decreased or held if needed due to adverse effects.
  Other Names: Jakavi

SUMMARY:
Alopecia areata (AA) is a common disease of the immune system, known as an "autoimmune" disease. In the disease, the immune system mistakenly destroys the hair follicle, causing hair to fall out. Despite many people having this disease, research into its cause and into new, better ways to treat AA has lagged far behind other similar diseases of the immune system. Currently, there are no Federal Drug Administration approved drugs for AA.

Ruxolitinib (made by Incyte) is an intervention known to effectively treat a disease of the bone marrow, known as myelofibrosis. It is also being studied in the treatment of rheumatoid arthritis, another "autoimmune" disease, by fighting inflammation. There are some genetic and chemical similarities between those with myelofibrosis, active rheumatoid arthritis and AA, suggesting that treatment with ruxolitinib may be effective in AA. In mice specially designed for testing drugs for the treatment of human alopecia areata, this medication worked to prevent the disease AA from starting in mice that would have otherwise developed the disease. To test Ruxolitinib, we are going to treat 12 patients with moderate to severe AA for a minimum of 3 months up to 6 months. This is an "open-label" study, meaning that there will not be a placebo group; all patients enrolled in the study will receive the active medication. The effectiveness of the medication will be measured by changes in hair re-growth as determined by physical exam and photography, as well as by patient and physician scoring. Patients will be followed for another 3 months off of the drug to see if the effects of treatment last and if there is delayed response. The safety of the medication, ruxolitinib, in patients with alopecia areata will also be evaluated.

Blood work will be collected before medication is started, during the treatment period, and after ruxolitinib is stopped, in order to monitor for adverse effects of the medication. Small scalp biopsies and peripheral blood will be taken at the beginning of the study before treatment and also after 12 and possibly 24 weeks. Optional biopsies may also be taken at additional time points based on clinical considerations. The chemical analysis of these skin samples and blood will help us to understand how the disease happens, how the treatment works, and may even guide us to better treatments in the future.

DETAILED DESCRIPTION:
Alopecia areata (AA) is a common autoimmune disease resulting from immune destruction of the hair follicle and subsequent hair loss. Despite its high prevalence, research into the pathogenesis and the development of innovative therapies in AA has lagged far behind other autoimmune diseases. Currently, there are no FDA approved drugs for AA. Ruxolitinib (Incyte) is an intervention known to effectively treat myelofibrosis and also rheumatoid arthritis by modulating the inflammatory response of the interferon response pathway by inhibition of Jak1/Jak2. Rheumatoid arthritis shares several susceptibility genes in common with AA. All three diseases share the central role of the interferon-gamma response pathway, which is the rationale for selecting Ruxolitinib for evaluation in this clinical trial. Both systemic and topical Ruxolitinib have been shown to prevent the onset of AA in the C3H-HeJ animal model of AA, demonstrating preclinical proof-of-concept data in AA. To test the safety and efficacy of Ruxolitinib in patients with moderate to severe AA, we propose this open-label, single arm pilot study with a total of 12 patients, treated for a minimum of 3 months up to 6 months. Efficacy will be measured by changes in hair re-growth as determined by physical exam and photography, as well as by patient and physician global evaluation scores. Patients will be followed for another 3 months to evaluate durability of response following the treatment phase. Punch biopsies and peripheral blood will be obtained at baseline prior to treatment and then after 12 and possibly 24 weeks for immune monitoring and for molecular studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 75 years of age.
* Patients with a diagnosis of patch type alopecia areata.
* Patients will have >30% and <95% total scalp hair loss at baseline as measured using the SALT score. Two patients with current episodes of alopecia totalis/universalis may be included in this study.
* Duration of hair loss greater than 3 months.
* No evidence of regrowth present at baseline.
* Patients may be naïve to treatment or unresponsive to intralesional (IL) steroids or other treatments for alopecia areata.

Exclusion Criteria:

* Patients with a history of or active skin disease on the scalp such as psoriasis or seborrheic dermatitis.
* Patients in whom the diagnosis of alopecia areata is in question.
* Patients with active medical conditions or malignancies (except adequately treated basal or squamous cell carcinoma) that in the opinion of the investigator would increase the risks associated with study participation, including patients with a history of recurrent infections.
* Women of childbearing potential who are unable or unwilling to use two forms of birth control for the study duration.
* Women who are pregnant or nursing.
* Patients known to be HIV or hepatitis B or C positive.
* Patients with history or evidence of hematopoietic abnormality.
* Patients with <200K platelet count at baseline.
* Patients with history or evidence of renal or hepatic impairment.
* Patients with history of immunosuppression or history of recurrent serious infections.
* Patients unwilling or unable to discontinue treatments known to affect hair regrowth in AA.
* Patients taking any medication considered a strong CYP3A4 inhibitor who is unable or unwilling to stop this medication for the duration of the study.
* Patients receiving treatment deemed to affect alopecia areata within 2 weeks to one month of baseline visit depending on the specific treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Mackay-Wiggan, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, Department of Dermatology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mackay-Wiggan J, Jabbari A, Nguyen N, Cerise JE, Clark C, Ulerio G, Furniss M, Vaughan R, Christiano AM, Clynes R. Oral ruxolitinib induces hair regrowth in patients with moderate-to-severe alopecia areata. JCI Insight. 2016 Sep 22;1(15):e89790. doi: 10.1172/jci.insight.89790. PMID 27699253

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in SALT Score
Description: Severity of Alopecia Tool Score (SALT) calculation is based on a scoring system. The scalp is divided into the following 4 areas: 1) Vertex: 40% (0.4) of scalp surface area, 2) Right profile of scalp: 18% (0.18) of scalp surface area, 3) Left profile of scalp: 18% (0.18) of scalp surface area, and 4) Posterior aspect of scalp: 24% (0.24) of scalp surface area. The percentage of hair loss in any of these areas is the percentage hair loss multiplied by percent surface area of the scalp in that area. The SALT score is the sum of percentage of hair loss in all the above-mentioned areas, so a lower number indicates a better outcome. The reported SALT score range is from a minimum of 0 (no hair loss) to a maximum of 100 (100% hair loss).
Time Frame: Baseline, 3 months and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 12
score on a scale
  Baseline | 65.8 (28.0)
  3 months | 24.8 (22.9)
  6 months | 7.3 (13.5)

2. Secondary Outcome: Percentage of Regrowth
Description: Mean percentage of regrowth was calculated at the end of treatment for all subjects.
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: percentage of regrowth
Groups:
- Ruxolitinib: A fixed dose of ruxolitinib (20mg) will be self-administered orally twice daily for 12 to 24 weeks. Dosing may be decreased or held if needed due to adverse effects.
  Ruxolitinib: A fixed dose of ruxolitinib (20mg) will be self-administered orally twice daily for 12 to 24 weeks. Dosing may be decreased or held if needed due to adverse effects.
  No serious adverse effects noted
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 12
percentage of regrowth | 68.9 (42.6)

ADVERSE EVENTS:
Time Frame: 9 months per patient
Arm/Group | Ruxolitinib
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib (N=12)
upper respiratory infection (Infections and infestations) | 5 (7)
low hemoglobin (Blood and lymphatic system disorders) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 2 (2)
pneumonia (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No